CLINICAL TRIAL: NCT05527171
Title: Virtual Reality Mindfulness Meditation in Patients After Anterior Cruciate Ligament Reconstruction
Brief Title: Virtual Reality Mindfulness Meditation After ACL Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-0493; K23AR079056 (NIH)
Record Dates: First submitted 2022-08-25; First posted 2022-09-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: Neurosciences; Rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Mindfulness Meditation Group (Experimental): Participants will complete 8-weeks of virtual reality mindfulness meditation and an advanced neuromuscular training program. Mindfulness meditation is the practice of sustaining attention on the body, breath, or sensations in any given moment and allows for the self-regulation of attention by decreasing rumination about past or future events. During the practice of mindfulness meditation, the individual is aware of all incoming thoughts and feelings, but rather than reacting to them, the individual accepts them. Virtual reality mindfulness meditation has been demonstrated to be superior in inducing mindfulness states when compared to traditional mindfulness meditation. Use of a virtual reality system to implement mindfulness meditation not only decreases the barrier of time to implement psychological interventions, but also improves the clinician's confidence in implementing the intervention as the virtual reality system guides the patient through the mindfulness meditation process.
  Interventions: Behavioral: Virtual Reality Mindfulness Meditation
- VR Sham Group (Sham Comparator): Participants will complete 8-weeks of virtual reality sham and an advanced neuromuscular training program. Participants will be immersed in a virtual environment but will not receive the mindfulness meditation.
  Interventions: Behavioral: Virtual Reality Sham

INTERVENTIONS:
Behavioral: Virtual Reality Mindfulness Meditation — Participants will be immersed in a virtual environment of their choosing. While in the virtual environment, participants will follow a guided mindfulness meditation script. Participants will complete the intervention 3 times a week over the course of 8-weeks.
  Arms: VR Mindfulness Meditation Group
Behavioral: Virtual Reality Sham — Participants will be immersed in a virtual environment of their choosing, such as at a beach, forest, or lake.
  Arms: VR Sham Group

SUMMARY:
To evaluate the effect of virtual reality mindfulness meditation on patients after ACLR, the investigators will determine the effect of virtual reality mindfulness meditation to 1) decrease self-reported injury-related fear, 2) improve poor jump-landing movement patterns, and 3) improve brain activity in women 1 to 5 years post-ACLR when compared to a virtual reality sham group.

DETAILED DESCRIPTION:
Injury-related fear after anterior cruciate ligament (ACL) injury significantly contributes to decreased return to sport, decreased physical activity engagement, and increased ACL reinjury risk in previously high functioning, physically active individuals. Injury-related fear is also associated with poor jump-landing movement patterns in patients after ACL reconstruction (ACLR). Unfortunately, current rehabilitation practices do not specifically address injury-related fear in patients after ACLR. Virtual reality mindfulness meditation is a mental practice that involves focusing the mind on experiences in the present moment and has been used to address depression, anxiety, and chronic musculoskeletal pain. To evaluate the effect of virtual reality mindfulness meditation on patients after ACLR, the investigators will determine the effect of virtual reality mindfulness meditation to 1) decrease self-reported injury-related fear, 2) improve poor jump-landing movement patterns, and 3) improve brain activity in women 6 months to 10 years post-ACLR when compared to a virtual reality sham group. Patients in the intervention group will complete 8-weeks of virtual reality mindfulness meditation + an advanced rehabilitation training program. Patients in the sham group will complete 8-weeks of the virtual reality sham + an advanced rehabilitation training program. The central hypothesis is that women 6 months to 10 years post ACLR who undergo virtual reality mindfulness meditation will demonstrate decreased injury-related fear, improved jump-landing movement patterns, and improved brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 14-25 years
* Have self-reported levels of fear on the Tampa Scale of Kinesiophobia-11
* Have poor jump-landing movement quality as measured by the Landing Error Scoring System-Real Time
* Injured their knee playing or training for sports (recreational or organized)
* Right-hand dominant
* 6 months to 10-years post-ACLR
* Demonstrate magnetic resonance imaging (MRI) compliance

Exclusion Criteria:

* Male
* Concussion in the past 3 months
* Presence of metal fragments, pins, plates, or clips, shrapnel, permanent makeup, body piercings that cannot be removed, surgical implants, or orthodontics that cannot be removed
* On any medication that affects the central nervous system
* Any neurological conditions (i.e. epilepsy)
* Claustrophobia
* Under the influence of alcohol or other recreational drugs
* Pregnancy or suspicion of pregnancy

Ages: 14 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who were eligible and enrolled in the study | Through study completion, a total of approximately 3 years.
  Feasibility of the Virtual Reality and Advanced Neuromuscular Training Rehabilitation Program will be assessed through established recruitment for patients post-ACLR. Recruitment is defined as the percentage of participants who were eligible and enrolled in the study.
Percentage of participants retained in the study | Through study completion, a total of approximately 8-weeks
  Feasibility of Virtual Reality and Advanced Neuromuscular Training Rehabilitation Program will be assessed to determine participant retention. Retention is defined as the percentage of participants enrolled and who have completed all study measures through 8-weeks.
Mean Acceptability Survey Score | Collected post-treatment after completion of the intervention/sham at week 8
  Feasibility of Virtual Reality and Advanced Neuromuscular Training Rehabilitation Program will be assessed via an acceptability survey during the final assessment post-treatment at week 8. Mean score greater than 8 will be interpreted as high acceptability.
Change in Injury-related fear as measured by the Tampa Scale of Kinesiophobia-11 | Collected at baseline and post-treatment after completion of the intervention/sham at week 8
  The Tampa Scale of Kinesiophobia-11 is a patient-reported outcome measure that assesses fear of movement and/or reinjury. This is an 11-item questionnaire that is valid. Scores range from 11 to 44, with higher scores indicating elevated fear.

SECONDARY OUTCOMES:
Change in external knee abduction moment | Collected at baseline and post-treatment after completion of the intervention/sham at week 8
  External knee abduction moment is a biomechanical assessment pertinent to patients with ACL reconstruction. Increased knee abduction moment has been associated with ACL reinjury risk. Patients will complete a jump-landing task to assess knee abduction moment using a three-dimensional motion capture system and embedded force plates.
Change in knee flexion excursion | Collected at baseline and post-treatment after completion of the intervention/sham at week 8
  Knee flexion excursion is a biomechanical assessment pertinent to patients with ACL reconstruction. Decreased knee flexion excursion has been associated with ACL reinjury risk. Patients will complete a jump-landing task to assess knee flexion excursion using a three-dimensional motion capture system and embedded force plates.
Change in Mean percent Blood Oxygen Level Dependent signal in Default Mode Network. | Collected at baseline and post-treatment after completion of the intervention/sham at week 8
  Blood Oxygen Level Dependent (BOLD) fMRI is a non-invasive diagnostic method of assessing brain activity by detecting signal changes secondary to changes in blood flow and oxygenation. Increased mean percent BOLD signal is associated with increased brain activity and decreased mean percent BOLD is associated with decreased brain activity.
  BOLD signal will be measured during a picture imagination task with sport-specific images and activity of daily living (ADL) images presented during the fMRI scan. Images are presented for 3 seconds with a 12-second rest between images. Whole brain functional images will be collected via a 3T PRI Scanner. Functional data will be acquired with BOLD echoplanar imaging (EPI) and processed using Analysis of Functional NeuroImages (AFNI). Mean BOLD percentage change based on image category, sport-specific versus ADL, will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Shelby E Baez, Ph.D., ATC, Principal Investigator — UNC-Chapel Hill
Locations (1):
- Fetzer Hall, 210 South Road, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from all patients regardless of successful completion of the proposed experimental protocol; except if a patient/guardian withdraws their consent. The final dataset will include demographic information, self-reported knee function and injury-related fear questionnaires, biomechanics analysis summaries and raw functional magnetic resonance imaging data. Accompanying the data, a documentation file will be provided containing the methodological procedures used during the collection of the data and providing a key for all variables included within the final dataset. Prior to sharing this data, all personal identifying information will be removed to protect the rights and privacy of the patients.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication.
Access Criteria: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
  To further protect the privacy and confidentiality of the data, the data and associated documentation will be made available only under a data-sharing agreement that provides for: (1) requirements to protect patients' privacy and data confidentiality including appropriate data security; (2) restrictions for the transferring of data to others; (3) commitments that the data will be used for research purposes only and not for a profit-making enterprise, and (4) prohibition of manipulation of data for the purposes of attempting to identify research participants.